CLINICAL TRIAL: NCT00875316
Title: A Randomised, Double-blind, Multiple Dose-ascending, Placebo-controlled Study in Healthy Volunteers and Parkinson's Disease Patients to Assess the Safety, Tolerability and PK of Daily Oral Administration of Cogane™ Over One Month
Brief Title: Safety and Tolerability Study of Cogane™ in Healthy Volunteers and Parkinson's Disease Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Phytopharm (Industry)
Responsible Party: Mrs. Joanna Locker, Phytopharm plc
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P58/07CL/ST/08/01; LCG 2237/08
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Phase I
MeSH Terms: conditions — Parkinson Disease | interventions — sarsasapogenin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort A (Experimental)
  Interventions: Drug: Cogane™ (PYM50028)
- Cohort B (Experimental)
  Interventions: Drug: Cogane™ (PYM50028)
- Cohort C (Experimental)
  Interventions: Drug: Cogane™ (PYM50028)
- Cohort D (Optional) (Experimental)
  Interventions: Drug: Cogane™ (PYM50028)

INTERVENTIONS:
Drug: Cogane™ (PYM50028) — Orally active neurotrophic factor inducer

SUMMARY:
Phytopharm plc is developing Cogane™ which is a new medicine for the treatment of Parkinson's disease (PD). The purpose of the study is to find out if Cogane is safe and well tolerated in both healthy volunteers and Parkinson's disease patients and to determine if there is a difference in the way that the body deals with Cogane (pharmacokinetics) between these two groups.

It is expected that the study will prove that Cogane™ is safe and well tolerated and will provide us with a pharmacokinetic profile for both subject groups.

ELIGIBILITY:
Key Inclusion Criteria (Healthy Volunteers):

* Male & Female healthy volunteers aged between 40 and 80 years at the time of informed consent
* Females of non-childbearing potential
* General Good Health

Key Exclusion Criteria (Healthy Volunteers):

* No clinically significant and relevant medical history
* Smoked within the 3 months prior to screening
* Use of prescription or non-prescription systemic or topical medication (including herbal remedies) within 14 days of the first dose administration

Key Inclusion Criteria (Parkinson's disease patients):

* Male & Female Parkinson's disease patients aged between 40 and 80 years at the time of informed consent
* Must have a diagnosis of idiopathic Parkinson's disease according to the UK Parkinson's Disease Society Brain Bank criteria
* Subjects who are taking Parkinson's disease treatments should be on a stable regimen for at least 4 weeks prior to screening

Key Exclusion Criteria (Parkinson's disease patients):

* Diagnosis of dementia
* Parkinson's disease of a known genetic cause
* History of surgical intervention for Parkinson's disease

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of Cogane™ oral solution | Throughout 28 day dosing period

SECONDARY OUTCOMES:
To investigate the pharmacokinetic profile of Cogane™ and its metabolites | Throughout 28 day dosing period

CONTACTS AND LOCATIONS:
Overall Officials: Investigator, Principal Investigator — Cambridge, UK
Locations (1):
- LCG Bioscience, Bourn, Cambridgeshire, United Kingdom